CLINICAL TRIAL: NCT04249518
Title: Video Extradition of Continuous Positive Airway Pressure - Influence on Compliance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15022020
Record Dates: First submitted 2020-01-17; First posted 2020-01-31 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-10

CONDITIONS: Patient Empowerment; Patient Engagement; Patient Compliance
MeSH Terms: conditions — Patient Participation; Patient Compliance

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nurse instruction of CPAP (No Intervention): Normal extradition. 45 minutes face to face with a nurse.
- Video extradition (Experimental): Access to 7 min video - explaining how to start CPAP and how to adjust the mask.
  Interventions: Behavioral: Videoeducation

INTERVENTIONS:
Behavioral: Videoeducation — No drugs used. The only difference in the to arms is the way the extradition is.
  Arms: Video extradition

SUMMARY:
Confirming or denying it in the future is an opportunity for certain patient groups to have the option of video delivery. So that in calm circumstances and possibly. several times can review the video and equipment in the home and hopefully achieve the same or better compliance with the ongoing treatment.

DETAILED DESCRIPTION:
Due to increasing age, BMI and increased focus on obstructive sleep apnea syndrome (OSAS) in the background population, an increasing number of obstructive sleep apnea (OSA) patients are expected to occur in the coming years. This is accompanied by a need for multiple deliveries of CPAP equipment, which is the recommended treatment. A large proportion of patients are young and healthy with their OSA. There is an increased focus on telemedicine and much of the control of patients has been transferred to ambuflex, where treatment effect or treatment problems can be more easily detected. Socioeconomically, the deliveries, together with the medical examination, are resource-intensive and they also take up a lot of the patient's time and often at distant times. The quality of disclosure and information varies greatly in both time and amount of information. The large amount of information can be difficult to remember for patients and relatives. Most investigations require more visits to the hospital and therefore potentially provide several days away from work.

A similar trial has never been made, but randomized studies have been made in the past where the delivery of CPAP or low compliance patients has been supported by a motivational video or teaching with good effect. Studies have also been conducted that have attempted to identify CPAP dropout and compliance based on gender, age, educational level and personality, with unemployment being the only contributing prognostic factor in the negative direction. It is well-studied that if patients suffer from insomnia, the onset of CPAP can be difficult and this patient group should be monitored more closely and possibly. have additional help for startup.

The video in this study provides a brief review of illness and treatment, instruction on assembling and adapting equipment, and answers to the most frequently asked questions. Both groups are given the same telephone numbers as usual, for questions and here it will be included in the study if there is a difference in the amount of contacts to the ambulatory. The video has been tested in the relevant setting before starting the project. M Gaglianos made in 1988 is a literature review showing that video teaching is good and more effective than traditional teaching methods, with effects on short-term but not long-term memory.

ELIGIBILITY:
Inclusion Criteria:

* candidate to CPAP
* over age of 18

Exclusion Criteria:

* Language issues
* sight or hearing handicap
* kognitive issues
* if drivers license is confiscated

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1234 (Estimated)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2022-02-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
compliance in percentage | one month.
  Compliance at one month follow up. Minimum 0 % maximum 100 % compliance.

SECONDARY OUTCOMES:
Depression | one month.
  Depression measured by major depression index (MDI) questionnaire.MDI total score < 20 being normal and not depressed. MDI total score > 29 indicating severe depression.
Influencer | one month.
  Education level registered by ISCED 2011 levels of education. Level 0-8. 8 being doctoral or equivalent. 0 being Early childhood Education (01 Early childhood educational development)
Insomnia | One month .
  Insomnia measured by insomnia severity index (questionnaire). 0-12 points. 0 being no problems facing a sleep. 12 having lots og trouble falling a sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Bille, MD, Principal Investigator — University Aarhus

IPD SHARING:
Plan to Share IPD: No